CLINICAL TRIAL: NCT05122403
Title: Multimodal Magnetic Resonance Imaging Study for Magnetic Resonance-Guided Focused Ultrasound Central Lateral Thalamotomy in Neuropathic Pain
Brief Title: Multimodal MRI for MRgFUS Central Lateral Thalamotomy in Neuropathic Pain
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Deputy Director of Department of Radiology, Chinese PLA General Hospital
Other Study IDs: MRgFUS-CL Neuropathic Pain
Record Dates: First submitted 2021-07-31; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Neuropathic Pain; Magnetic Resonance Imaging
Keywords: MR-guided focused ultrasound; Central Lateral Nucleus of Thalamus
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FUS Thalamotomy: The cohort includes patients with neuropathic pain who underwent MRgFUS central lateral thalamotomy.
  Interventions: Procedure: MRgFUS central lateral thalamotomy
- Sham Procedure: The cohort includes patients with neuropathic pain who underwent sham MRgFUS central lateral thalamotomy.

INTERVENTIONS:
Procedure: MRgFUS central lateral thalamotomy — MRgFUS central lateral thalamotomy is a minimally invasive and effective procedure for medication-refractory neuropathic pain patients.
  Groups: FUS Thalamotomy

SUMMARY:
To explore the pathogenesis underlying neuropathic pain as well as the mechanisms of pain relief after Magnetic resonance-guided focused ultrasound (MRgFUS) Central Lateral Thalamotomy through multi-model MRI study, and to identify imaging biomarkers for triaging patients and predicting the clinical outcomes. Craniofacial neuropathic pain is one of the most serious debilitating symptoms, leading to emotional disorders and poor quality of life. Previous studies have shown that Magnetic resonance-guided focused ultrasound (MRgFUS) central lateral thalamotomy is a minimally invasive and effective procedure for medication-refractory neuropathic pain patients. However, the clinical benefits were variable among individuals. It is important to clarify the pathogenesis of neuropathic pain and the mechanisms of pain relief induced by MRgFUS central lateral thalamotomy to triage suitable candidates for the procedure and predict clinical outcomes. In addition, localization precision and individualized treatment remain to be improved.

DETAILED DESCRIPTION:
The study was designed as a prospective, sham-controlled randomized clinical trial (randomized 1:1) with double-blinded assessments through the 3-month primary end point analysis. Patients assigned to a sham procedure were offered open label treatment after the 3-month blinded assessment. All treated patients were followed unblinded to 1 year. Baseline clinical demographics, Numerical Pain Rating Scale (NPRS) treatment parameters (energy, power, duration time, temperature, target location) , associated adverse effects were recorded

Imaging protocols:

T2; T2 Flair; DWI; ESWAN; MRS; 3D ASL 2.0s; 3D-T1; DTI; rs-functional MRI

Imaging evaluation:

1. Lesion appearance and volume are measured by T2, T2 Flair, DWI, ESWAN, 3D-T1;
2. ESWAN and MRS manifests the changes of iron deposition and metabolism, respectively;
3. ASL shows regional cerebral blood flow associated with the procedure;
4. DTI demonstrates the destruction of white matter integrity.
5. Rs-functional MRI reflects alterations of resting-state brain activity.

Treatment:

MRgFUS central lateral thalamotomy

Follow-up:

MRI + clinical evaluation：Baseline, 3-day, 1-month, 3-months, 6-months,12-months

ELIGIBILITY:
Inclusion Criteria:

1. Male and female, aged between 18 and 75 (inclusive);
2. Subjects who are able and willing to participate in the study;
3. Chronic neuropathic pain with disease duration lasting more than 6 months;
4. The worst NPRS score was ≥ 5 (out of 10), and the subjects reported a similar degree of pain in at least the past two months;
5. Medication-refractory neuropathic pain with resistance to at least three kinds of neuropathic pain prescription drugs and one interventional procedure

Exclusion Criteria:

1. Craniofacial pain syndrome associated with malignant tumors of the head and neck;
2. Idiopathic trigeminal neuralgia;
3. Headache syndrome, such as migraine;
4. Temporomandibular joint syndrome;
5. Atypical facial pain or pain related to somatoform disorders;
6. Subjects are regarded as unqualified candidates by experts;
7. active mental illness;
8. unstable heart state;
9. severe hypertension (diastolic blood pressure after taking medicine >100mm/Hg)
10. MR imaging standard contraindications, such as non-MRI compatible implanted metal devices, including pacemakers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic Neuropathic Pain
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-08-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
primary efficacy outcome（Numerical Pain Rating Scale score） | 1 years
  The primary efficacy outcome was determined by comparing the change from baseline to 3 months in the NPRS (Numerical Pain Rating Scale) score between FUS thalamotomy and sham procedures using intention-to-treat analysis.
Primary safety outcome（incidence and severity of adverse events） | 1 years
  Primary safety outcome was assessed by monitoring the incidence and severity of the procedure-related adverse events from the procedure through 1 year after treatment for all patients

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lou, MD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided